CLINICAL TRIAL: NCT07018388
Title: Intrapatient Comparison of Subthalamic and Globus Pallidus Internus Temporal Interference Stimulation in Parkinson's Disease
Brief Title: Intrapatient Comparison of STN and GPi tTIS in PD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025140B
Record Dates: First submitted 2025-06-05; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: subthalamic nucleus; Globus Pallidus Internus; transcranial temporal interference stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STN-tTIS (Experimental): Patients in this group receive 20 minutes of individualized 130 Hz STN-tTIS sessions targeting the more affected hemisphere's STN during medication "on" and are evaluated for the MDS-UPDRS-Ⅲ before and after treatment.
  Interventions: Device: NervioX-2400
- GPi-tTIS (Experimental): Patients in this group receive 20 minutes of individualized 130 Hz GPi-tTIS sessions targeting the more affected hemisphere's STN during medication "on" and are evaluated for the MDS-UPDRS-Ⅲ both before and after treatment.
  Interventions: Device: NervioX-2400

INTERVENTIONS:
Device: NervioX-2400 — To design the individualized STN-tTIS, each patient completes a T1-weighted anatomical magnetic resonance imaging (MRI) scan. The individual's structural brain MRI data are used to determine the STN-tTIS montage and stimulation settings through computational modeling.
  Arms: GPi-tTIS
Device: NervioX-2400 — To design the individualized GPi-tTIS, each patient completes a T1-weighted anatomical magnetic resonance imaging (MRI) scan. The individual's structural brain MRI data is used to determine the GPi-tTIS montage and stimulation settings via computational modeling.
  Arms: STN-tTIS

SUMMARY:
The goal of this clinical trial is to evaluate the immediate effects and conduct intrapatient comparisons of individualized 130 Hz Subthalamic Nucleus-transcranial Temporal Interference Stimulation (STN-tTIS) and Globus Pallidus Internus-transcranial Temporal Interference Stimulation (GPi-tTIS) on motor symptoms in patients with early to mid-stage Parkinson's Disease (PD) during "on" medication states.

The main questions this study aims to answer are:

1. Is the therapeutic effect of STN-tTIS superior to that of GPi-tTIS?
2. What is the degree of improvement in motor symptoms of Parkinson's Disease patients after receiving STN-tTIS or GPi-tTIS during the "on" medication phase?

Researchers will compare the MDS-UPDRS-III improvement scores of tTIS therapy at different targets. Participants are required to:

1. Visit the clinic twice within two weeks for therapy and testing.
2. Record their symptoms and scores.

DETAILED DESCRIPTION:
This clinical trial aims to explore which targets are better for improving PD motor symptoms. Patients were randomly assigned to either Group A or Group B. Group A first received STN-tTIS therapy, followed by GPi-tTIS therapy; Group B received the treatments in the reverse order. Each session lasted 20 minutes, and patients were in the on-medication state for both treatments. The order of sessions was randomized, with at least 7 days of washout between sessions to avoid carryover effects. MDS-UPDRS-III evaluations were assessed before and after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Parkinson's disease (MDS);
* Hoehn & Yahr stage < 3;
* Antiparkinsonian drugs must have remained unchanged in the past four weeks, and the dosage must have remained stable throughout the study.

Exclusion Criteria:

* Presence of neurological disorders that may affect the study (e.g., traumatic brain injury);
* History of antipsychotics, antidepressants, or dopamine modulators outside of PD drugs;
* Metal devices in the head or heart (e.g., deep brain stimulators, pacemakers);
* Unstable vital signs.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS-Ⅲ scores | pre-intervention, immediately after the intervention
  The score range for MDS-UPDRS-III is from 0 to 132. The minimum value is 0, indicating no motor impairment, and the maximum value is 132, indicating the most severe motor impairment. Higher scores on the MDS-UPDRS-III indicate worse outcomes, as they reflect greater severity of motor symptoms.

SECONDARY OUTCOMES:
MDS-UPDRS-Ⅲ sub-scores | pre-intervention, immediately after the intervention
  The MDS-UPDRS-III assesses motor symptoms in Parkinson's disease through sub-scores: Tremor Sub-score: Items 15-18; range 0-16. Higher scores indicate more severe tremors. Rigidity Sub-score: Item 3; range 0-12. Higher scores reflect greater rigidity. Bradykinesia Sub-score: Items 2, 4-9, and 14; range 0-40. Higher scores indicate more severe slowness of movement. Axial Sub-score: Items 1 and 9-13; range 0-24. Higher scores suggest more significant axial impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No